CLINICAL TRIAL: NCT06756945
Title: Low-dose Evaluation of Aspirin After STEMI Patients With PCI: A Multicenter, Double-blind, Randomized Controlled Clinical Trial
Acronym: LEAST
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024AZB1004; 2024AZB1004 (Other Grant/Funding Number: Beijing Anzhen Hospital High Level Research Funding)
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: ST-elevation Myocardial Infarction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin 50mg/d (Experimental): STEMI patients receive aspirin 50 mg once daily (one 50 mg aspirin tablet plus one matching placebo tablet) plus ticagrelor 90 mg twice daily
  Interventions: Drug: aspirin 50 mg once daily (one 50 mg aspirin tablet plus one matching placebo tablet) plus ticagrelor 90 mg twice daily
- Aspirin 100mg/d (Active Comparator): STEMI patients receive aspirin 100 mg once daily (two 50 mg aspirin tablets) plus ticagrelor 90 mg twice daily
  Interventions: Drug: aspirin 100 mg once daily (two 50 mg aspirin tablets) plus ticagrelor 90 mg twice daily

INTERVENTIONS:
Drug: aspirin 50 mg once daily (one 50 mg aspirin tablet plus one matching placebo tablet) plus ticagrelor 90 mg twice daily — STEMI patients receive aspirin 50 mg once daily (one 50 mg aspirin tablet plus one matching placebo tablet) plus ticagrelor 90 mg twice daily
  Arms: Aspirin 50mg/d
Drug: aspirin 100 mg once daily (two 50 mg aspirin tablets) plus ticagrelor 90 mg twice daily — STEMI patients receive aspirin 100 mg once daily (two 50 mg aspirin tablets) plus ticagrelor 90 mg twice daily
  Arms: Aspirin 100mg/d

SUMMARY:
The study aims to optimize the dual antiplatelet therapy regimen for patients with STEMI after PCI, focusing on addressing the following key technical challenges: establishing an effectiveness evaluation system for a low-dose aspirin (50mg/day) antithrombotic treatment strategy based on ticagrelor, including the formulation of a scientific non-inferiority margin, assessment criteria, and composite endpoint determination standards; constructing a strict risk assessment system for major bleeding events, including bleeding event grading based on BARC standards and a blind evaluation process by an independent endpoint event adjudication committee; and developing a quality control system for multicenter clinical research to ensure patient follow-up compliance and data reliability. By solving the above technical challenges, the study provides evidence-based medical support and technical support for optimizing the antithrombotic treatment regimen for STEMI patients after PCI.

ELIGIBILITY:
Inclusion Criteria:

STEMI patients with clear diagnosis Has received PCI treatment (at least the culprit's blood vessels have been treated); 18 years old and above, regardless of gender; Received DAPT upon discharge: aspirin+ticagrelor; Signed informed consent form approved by the ethics committee

Exclusion Criteria:

Individuals with atrial fibrillation/DVT/valve surgery requiring anticoagulant medication; Combined cardiomyopathy (HCM/DCM/RCM); Combining severe ventricular arrhythmias requires ICD; Chronic obstructive pulmonary disease (bronchial asthma, chronic bronchitis, emphysema, pulmonary heart disease); Serious infectious diseases, including active hepatitis B, hepatitis C or AIDS patients; Diseases of the blood system, such as thrombocytopenia, severe anemia, leukemia, etc; Severe liver and kidney dysfunction; Malignant tumors; Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3612 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint 1 (composite ischemic events for non-inferiority testing) | 12 months
  Primary Endpoint 1 (composite ischemic events for non-inferiority testing) includes all-cause death, non-fatal myocardial infarction, non-fatal stroke, and urgent/ischemia-driven target vessel revascularization
Primary Endpoint 2 (bleeding events for superiority testing) | 12 months
  Secondary endpoints at 12 months include individual components of the composite ischemic endpoint, stent thrombosis, and safety endpoints comprising BARC type 2-5 bleeding events, GUSTO mild, moderate, and severe/life-threatening bleeding, and non-CABG-related minimal, minor, and major bleeding

REFERENCES:
- [Derived] Zheng W, Gong ZT, Qian HY. Study protocol for low-dose evaluation of aspirin in patients with ST-elevation myocardial infarction undergoing percutaneous coronary intervention (LEAST): a multicenter, double-blind, randomized controlled clinical trial. Ann Med. 2025 Dec;57(1):2589577. doi: 10.1080/07853890.2025.2589577. Epub 2025 Nov 23. PMID 41277137